CLINICAL TRIAL: NCT04136873
Title: A Phase 1B Trial To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of CVL-231 in Subjects With Schizophrenia
Brief Title: A Multiple Ascending Dose Trial of CVL-231 in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CVL-231-SCH-001
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part A: 5 mg QD CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part A: 5 mg QD Placebo (Placebo Comparator): Matching Placebo; Oral Dose
  Interventions: Drug: Matching Placebo
- Part A: 10 mg QD CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part A: 10 mg QD Placebo (Placebo Comparator): Matching Placebo; Oral Dose
  Interventions: Drug: Matching Placebo
- Part A: 20 mg QD CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part A: 20 mg QD Placebo (Placebo Comparator): Matching Placebo; Oral Dose
  Interventions: Drug: Matching Placebo
- Part A: 5-10-20 mg BID CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part A: 5-10-20 mg BID Placebo (Placebo Comparator): Matching Placebo; Oral Dose
  Interventions: Drug: Matching Placebo
- Part A: 30 mg QD CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part A: 30 mg QD Placebo (Placebo Comparator): Matching Placebo; Oral Dose
  Interventions: Drug: Matching Placebo
- Part B 30 mg QD CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part B 30 mg QD Placebo (Placebo Comparator): Matching Placebo; Oral Dose
  Interventions: Drug: Matching Placebo
- Part B 20 mg BID CVL-231 (Active Comparator): Oral Dose
  Interventions: Drug: CVL-231
- Part B 20 mg BID Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: CVL-231 — CVL-231
  Arms: Part A: 10 mg QD CVL-231; Part A: 20 mg QD CVL-231; Part A: 30 mg QD CVL-231; Part A: 5 mg QD CVL-231; Part A: 5-10-20 mg BID CVL-231; Part B 20 mg BID CVL-231; Part B 30 mg QD CVL-231
Drug: Matching Placebo — Placebo matching CVL-231
  Arms: Part A: 10 mg QD Placebo; Part A: 20 mg QD Placebo; Part A: 30 mg QD Placebo; Part A: 5 mg QD Placebo; Part A: 5-10-20 mg BID Placebo; Part B 20 mg BID Placebo; Part B 30 mg QD Placebo

SUMMARY:
The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of CVL-231 following multiple-dose oral administration in subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a primary diagnosis of schizophrenia per DSM-5, as confirmed by the MINI.
2. Subjects with the following scores on the PANSS at time of signing ICF and at Day -1: • Positive Subscale 7 (hostility) ≤3 (normal to moderate) • General Psychopathology Subscale 8 (uncooperativeness) ≤3 (normal to moderate)
3. Subjects with the following scores (normal to mild symptoms) at time of signing ICF and at Day -1: • All individual items of the Modified SAS (M-SAS) <2 • All individual items (Items 1-7) of the Abnormal Involuntary Movement Scale (AIMS) <2 • Clinical global assessment item of the Barnes Akathisia Rating Scale (BARS) <3
4. Body mass index of 17.5 to 38.0 kg/m2 and a total body weight >50 kg (110 lbs).

Cohorts 1 Through 5 (Part A):

Subjects are eligible to be included in trial (Cohorts 1 through 5) only if all of the following additional criteria apply:

1. Male and female subjects, ages 18 to 50 years, inclusive.
2. Subjects with a score on the CGI-S ≤4 (normal to moderately ill) at time of signing ICF and at Day -1.
3. Subjects with a PANSS total score of ≤80 at the time of signing ICF and at Day -1.

Cohort 6 (Part B):

Subjects are eligible to be included in trial (Cohort 6) only if all of the following additional criteria apply:

1. Male and female subjects, ages 18 to 55 years, inclusive.
2. Subjects with a score on the CGI-S ≥4 (moderately to severely ill) at time of signing ICF and at Day -1.
3. Subjects with a PANSS total score of ≥80 at the time of signing ICF and at Day -1. Additionally, subjects must meet a score of ≥4 (moderate or greater) for ≥2 of the following Positive Scale items at the time of signing ICF and at Day -1:

   * Positive Scale 1 (delusions)
   * Positive Scale 2 (conceptual disorganization)
   * Positive Scale 3 (hallucinatory behavior)
   * Positive Scale 6 (suspiciousness/persecution)
4. Subjects with a history of relapse and/or exacerbation of symptoms when not receiving antipsychotic treatment, excluding the current episode.
5. Subjects must be experiencing an acute exacerbation or relapse of symptoms, with onset less than 2 months prior to signing ICF.

Exclusion Criteria:

1. Subjects with a current DSM-5 diagnosis other than schizophrenia including, but not limited to, mental retardation; schizoaffective disorder; schizophreniform disorder; psychotic depression; major depressive disorder; bipolar disorder; post-traumatic stress disorder; generalized anxiety disorder, obsessive compulsive disorder, eating disorders (bulimia, anorexia), or other anxiety disorders as a primary diagnosis (subjects with anxiety symptoms secondary to schizophrenia are allowed); delirium, dementia, amnestic, or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
2. Subjects with schizophrenia who were considered resistant/refractory to antipsychotic treatment by history or who had a history of failure to respond to clozapine or response to clozapine treatment only.
3. Subjects with EPS being treated with a medication that required dose modification and/or new treatment within 6 months prior to signing ICF.
4. Subjects with a current history of significant pulmonary, gastrointestinal, renal, hepatic, metabolic, endocrine (including newly diagnosed diabetes mellitus or subjects with known diabetes mellitus with glycosylated hemoglobin (HbA1c)>7.5%), hematological, immunological, psychiatric (excluding schizophrenia), or neurological disease.
5. Subjects with a current or past history of significant cardiovascular disease.
6. Subjects who experienced acute depressive symptoms within the past 30 days.
7. Subjects with epilepsy or a history of seizures, except for a single seizure episode, eg, a childhood febrile seizure, or a seizure related to trauma or alcohol withdrawal.
8. An active central nervous system infection, demyelinating disease, degenerative neurological disease, mental retardation, or any central nervous system disease deemed to be progressive.
9. History of moderate to severe substance or alcohol-use disorder (excluding nicotine or caffeine) as per DSM-5 criteria within 12 months prior to signing ICF.
10. Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent).
11. Human immunodeficiency virus seropositive status or acquired immunodeficiency syndrome, chronic hepatitis B or C.
12. Subject with a positive urine drug screen for illicit drugs or a positive breathalyzer test for alcohol.
13. Subjects with medically significant abnormal laboratory test results, vital sign results, or ECG findings.
14. Subjects who received transcranial magnetic stimulation or electroconvulsive therapy within 60 days of screening.
15. Any condition possibly affecting drug absorption, including bowel resections, bariatric weight loss surgery, or gastrectomy (this does not include gastric banding).
16. Subjects with difficulty swallowing.
17. Subjects with a history of neuroleptic malignant syndrome.
18. Subject who refuses to abstain from grapefruit-containing foods or beverages, or Seville orange-containing foods or beverages.

Cohorts 1 Through 5 (Part A) Subjects are excluded from the trial (Cohorts 1 through 5) if any of the following additional criteria apply:

1. Subjects who have experienced psychosis requiring hospitalization within the 6 months prior to signing ICF.
2. Subjects who experienced psychosis requiring a change in their antipsychotic medication (either drug type or dose) within the 3 months prior to signing ICF.
3. Subjects who fulfill any of the following dietary restrictions: • History of chronic consumption of >400 mg/day of caffeine-containing drinks or food • Refuses to abstain from caffeine-containing foods or caffeinated beverages for 48 hours prior to Day -1 through Follow up Visit • Refuses to abstain from alcohol from 7 days prior to Day -1 through Follow-up Visit
4. Subjects who have participated in any clinical trial within 60 days prior to signing ICF.
5. Subjects with a 12-lead ECG demonstrating any of the following:

   * Abnormal ST-T-wave morphologies that may interfere with QT analysis, such as flat or poorly defined end of the T wave or prominent U waves
   * Left ventricular hypertrophy
   * QT interval corrected for heart rate QTcF >450 msec
   * QRS interval >110 msec
   * Left or right bundle branch block
   * PR interval >240 msec
   * Heart rate <50 bpm or >90 bpm
   * Second- or third-degree atrioventricular block
6. Systolic blood pressure ≥130 mmHg and/or diastolic blood pressure ≥80 mmHg at Screening or Day -1, will be taken with subjects in the supine/semi-recumbent position, or symptomatic hypotension, or orthostatic hypotension, which is defined as a decrease of ≥20 mmHg in systolic blood pressure and/or a decrease of ≥10 mmHg in diastolic blood pressure after at least 3 minutes of standing compared with the immediately previous supine blood pressure. Subjects who are receiving chronic treatment with antihypertensive medications at Screening are also excluded.

Cohort 6 (Part B) Only Subjects are excluded from trial (Cohort 6 only) if any of the following additional criteria apply:

1. Subjects who have been hospitalized >14 days for the current episode of schizophrenia at the time of signing the ICF, excluding hospitalization for psychosocial reasons.
2. Subjects presenting with a first episode of schizophrenia, based on clinical judgment of the investigator.
3. Subjects with a 12-lead ECG exclusion as in Part A but will allow right bundle branch block in Part B.
4. Systolic blood pressure >130 mmHg and/or diastolic blood pressure >80 mmHg at Screening or Day -1 and subjects with orthostatic hypotension, defined as a decrease of ≥20 mmHg in systolic blood pressure and/or a decrease of ≥10 mmHg in diastolic blood pressure after at least 3 minutes of standing compared with the average resting supine/semi-recumbent blood pressure at Screening or Day -1, will be excluded. Subjects with a heart rate <50 bpm or >90 bpm. Subjects who are receiving chronic treatment with antihypertensive medications at Screening are also excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to Day 72
  Includes Incidence of Significant ECG Abnormalities Occurring Post-Baseline, significant changes in Vital signs (Systolic and Diastolic blood pressures, heart rate, respiratory rate and body temperature), and changes in laboratory measures (hematology, serum chemistry and urinalysis)
Incidence of suicidality as assessed by Columbia-Suicide Severity Rating Scale(C-SSRS) | Up to Day 72
  The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Change from Baseline of Simpson-Angus Scale (SAS) Results | Up to Day 72
  Evaluating Extrapyramidal symptoms using the SAS. The SAS consists of a list of 10 symptoms of parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms and a score of 4 representing a severe condition. The SAS total score is the sum of the scores for all 10 items.
Change from Baseline of Abnormal Involuntary Movement Scale (AIMS) Results | Up to Day 72
  The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Facial and oral movements (items 1 through 4), extremity movements (items 5 and 6), and trunk movements (item 7) are observed unobtrusively while the subject is at rest, and the investigator also makes global judgments on the subject's dyskinesias (items 8 through 10). Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, awareness, severe distress). In addition, the AIMS includes 2 yes/no questions that address the subject's dental status.
  The AIMS Movement Rating Score is defined as the sum of items 1 through 7 (ie, items 1 through 4, facial and oral movements; items 5 and 6, extremity movements; and item 7, trunk movements).
Change from Baseline of Barnes Akathisia Rating Scale (BARS) Results | Up to Day 72
  Evaluating Extrapyramidal symptoms using the BARS. The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the subject, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items are rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation is made on a 6-point scale, with a score of 0 representing absence of symptom and a score of 5 representing severe akathisia.

SECONDARY OUTCOMES:
Single-dose: Area under the plasma concentration vs. time curve (AUC) for CVL-231 and Metabolite (PF-06892787) | Day 1
Single-dose: Peak Plasma Concentration (Cmax) for CVL-231 and Metabolite (PF-06892787) | Day 1
Single-dose: Time to Maximum Concentration (Tmax) for CVL-231 and Metabolite (PF-06892787) | Day 1
Single-dose: Metabolite to parent ratio for Cmax for CVL-231 and Metabolite (PF-06892787) | Day 1
Single-dose: Metabolite to parent ratio for AUC tau for CVL-231 and Metabolite (PF-06892787) | Day 1
Multiple-dose: Steady state CVL-231 Peak Plasma Concentration (Cmax) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Time to Maximum Concentration (Tmax) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Trough plasma concentration (Ctrough) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Minimum blood plasma concentration (Cmin) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Area under the plasma concentration-time curve (AUCτ) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Area under the plasma concentration-time curve from time zero to infinity (AUCinf) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Apparent Total Clearance of Drug from plasma: CL/F for CVL-231 | Days 14 and/or 28 and/or 36
Multiple-dose: Steady-state average plasma drug concentration: Css for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Peak Trough Ratio (PTR) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Accumulation ratio calculated from Cmax,ss and Cmax after single dosing (Rac, Cmax) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Accumulation ratio calculated from AUCτ,ss and AUCτ after single dosing (Rac, AUC) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28 and/or 36
Multiple-dose: Elimination half-life (t½) for CVL-231 and Metabolite (PF-06892787) | Day 14-17 and/or Day 28-31
Multiple-dose: Elimination rate constant (kel) for CVL-231 and Metabolite (PF-06892787) | Day 14-17 and/or Day 28-31
Multiple-dose: Ae (amount eliminated unchanged in urine) for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28
Multiple-dose: Renal clearance for parent only for CVL-231 | Days 14 and/or 28
Multiple-dose: Metabolite to parent ratio for Cmax for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28
Multiple-dose: Metabolite to parent ratio for AUCtau for CVL-231 and Metabolite (PF-06892787) | Days 14 and/or 28

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, MD, Study Director — Cerevel Therapeutics, LLC
Locations (5):
- United States (5):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Woodlands International Research Group, Little Rock, Arkansas
  - Synergy San Diego, Lemon Grove, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Hassman Research Institute, Marlton, New Jersey

REFERENCES:
- [Derived] Krystal JH, Kane JM, Correll CU, Walling DP, Leoni M, Duvvuri S, Patel S, Chang I, Iredale P, Frohlich L, Versavel S, Perry P, Sanchez R, Renger J. Emraclidine, a novel positive allosteric modulator of cholinergic M4 receptors, for the treatment of schizophrenia: a two-part, randomised, double-blind, placebo-controlled, phase 1b trial. Lancet. 2022 Dec 17;400(10369):2210-2220. doi: 10.1016/S0140-6736(22)01990-0. PMID 36528376